CLINICAL TRIAL: NCT07004309
Title: Comparative Efficacy of Microfluidics and Density Gradient Centrifugation for Sperm Preparation in IVF: A Randomized Controlled Trial
Brief Title: Microfluidics Versus Density Gradient Centrifugation for Sperm Preparation in IVF
Acronym: MCvsDGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Do Thuy Huong, MD, PhD candidate, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-MCvsDGC-2025
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Male Infertility; Sperm DNA Fragmentation; In Vitro Fertilization (IVF)
Keywords: Microfluidics; Sperm DNA Fragmentation; In Vitro Fertilization; Sperm Preparation; ICSI
MeSH Terms: conditions — Infertility, Male | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel arms: microfluidic sperm sorting vs. density gradient centrifugation, with equal allocation.
Who Masked: Outcomes Assessor
Masking Description: Embryologists performing ICSI and embryo evaluation were blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microfluidics Group (Experimental): Semen samples are processed using a microfluidic sperm sorting device (ZyMot). Selected sperm are used for ICSI.
  Interventions: Procedure: Microfluidic sperm sorting
- DGC Group (Active Comparator): Sperm preparation using a discontinuous density gradient method with SpermGrad and SpermRinse media.
  Interventions: Procedure: Density Gradient Centrifugation

INTERVENTIONS:
Procedure: Microfluidic sperm sorting — Sperm selection using the ZyMot Microfluidic Sperm Separation Device. Process involves loading semen into microfluidic channels to isolate motile sperm with low DNA fragmentation.
  Arms: Microfluidics Group
Procedure: Density Gradient Centrifugation — Sperm preparation using a discontinuous density gradient technique with SpermGrad and SpermRinse media. Centrifugation separates motile sperm for use in ICSI.
  Arms: DGC Group

SUMMARY:
This randomized controlled trial aimed to compare the effectiveness of microfluidic sperm sorting and density gradient centrifugation (DGC) in reducing sperm DNA fragmentation index (DFI) and improving clinical outcomes in IVF. A total of 119 couples underwent IVF and were assigned to either microfluidic or DGC sperm preparation. The study evaluated sperm quality, fertilization, embryo development, and live birth rates.

DETAILED DESCRIPTION:
This single-center randomized controlled trial was conducted at Hanoi Medical University Hospital from March 2023 to March 2024. Couples undergoing IVF were randomized to two sperm preparation methods: microfluidics or density gradient centrifugation. Sperm DNA fragmentation index (DFI) was assessed before and after preparation. Primary outcomes included live birth rate and DFI reduction; secondary outcomes included sperm motility and morphology, fertilization rate, embryo quality, and pregnancy outcomes. The study received IRB approval and adhered to ethical standards.

ELIGIBILITY:
Inclusion Criteria:

* Female partner aged between 18 and 40 years
* Couples undergoing in vitro fertilization (IVF) cycles at the IVF and Tissue Engineering Center, Hanoi Medical University, between January 2022 and January 2024
* Use of autologous oocytes
* Use of ejaculated sperm
* Both partners provide written informed consent

Exclusion Criteria:

* Use of donor oocytes or donor sperm
* Requirement for testicular sperm extraction
* Diagnosis of oligoasthenozoospermia (OA) based on WHO 2021 criteria
* Female partner classified as having poor ovarian prognosis according to the POSEIDON 2016 criteria, including:

  * Anti-Müllerian hormone (AMH) level < 1.2 ng/mL
  * Antral follicle count (AFC) < 5
  * Or history of poor ovarian response (≤9 oocytes retrieved in previous cycles)
* Preimplantation genetic testing (PGT) cycles

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Sperm DNA Fragmentation Index (DFI) | Day of oocyte retrieval
  DFI measured before and after sperm preparation using SCSA method. Comparison between microfluidics and DGC groups
Live birth rate | Up to 9 months after embryo transfer
  Defined as the delivery of a live-born infant after 22 weeks of gestation. Comparison between microfluidics and DGC groups.

SECONDARY OUTCOMES:
Sperm motility after preparation | Immediately after sperm preparation
  Percentage of motile sperm, including both progressive and non-progressive motility, assessed post-preparation using WHO 2021 criteria.
Normal sperm morphology | Immediately after sperm preparation
  Percentage of sperm with normal morphology after preparation, assessed using strict WHO 2021 criteria.
Fertilization rate | 17-20 hours after ICSI
  Proportion of injected oocytes showing two pronuclei (2PN).
Good-quality embryo rate on Day 2 | Day 2 after fertilization
  Percentage of embryos with 4-6 blastomeres and <10% fragmentation on Day 2.
Biochemical pregnancy rate | 10-12 days after embryo transfer
  Defined as serum β-hCG >25 IU/L after embryo transfer.
Clinical pregnancy rate | 4 weeks after embryo transfer
  Presence of gestational sac and fetal heartbeat confirmed on ultrasound.
Ongoing pregnancy rate | 12 weeks after embryo transfer
  Viable intrauterine pregnancy confirmed by ultrasound at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Do Thuy Huong, PhD candidate, Principal Investigator — Hanoi Medical University
Locations (1):
- Center of IVF and Tissue Engineering, Hanoi Medical University Hospital, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of infertility treatment and to protect patient privacy in compliance with institutional ethics guidelines.